CLINICAL TRIAL: NCT05574452
Title: Specific Orientation in Anterior Cruciate Ligament Reconstruction: a Clinical Pilot Study
Brief Title: Patient Specific Instrumentation in ACL Reconstruction
Acronym: SONAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Medical Center Groningen (Other)
Collaborators: Ommelander Ziekenhuis Groningen (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 201400122
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: Patient specific instrumentation; ACL reconstruction; Femoral tunnel position
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Pilot Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pilot group (Experimental): Pilot group undergoing ACL reconstruction using the SONAR Femoral Aimer PSI
  Interventions: Device: ACL reconstruction using the SONAR Femoral Aimer PSI

INTERVENTIONS:
Device: ACL reconstruction using the SONAR Femoral Aimer PSI — ACL reconstruction using the SONAR Femoral Aimer PSI

SUMMARY:
Rationale: In anterior cruciate ligament (ACL) reconstruction, anatomical femoral tunnel positioning has proven to be difficult with current techniques. Limited visibility during surgery and high interpersonal variability are mainly responsible for non-anatomical femoral tunnel positioning. Non anatomical tunnel positioning can lead to long term failure of the reconstruction. In order to obtain an accurate and constant anatomical femoral tunnel position during ACL reconstruction, a patient specific surgical guide has been developed.

Objective: to assess the accuracy of the newly developed patient specific femoral aimer used during ACL reconstruction.

Study design: pilot study

Study population: 10 subjects (>16 years of age ) with ACL injury, requiring ACL reconstruction.

Intervention: all subjects will undergo ACL reconstruction in which a patient specific surgical guide is used for femoral tunnel positioning.

Main study parameters/endpoints: the main study parameter is the difference between the planned femoral tunnel position and the achieved tunnel position. This difference is quantified in both mm (translation) and degrees (rotation).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: No additional perioperative risks are associated with participation. Based on previous cadaver experiments, the accuracy of the patient specific, 3D printed femoral aimer is high. Subjects will undergo 1 postoperative MRI which will take place during a routine scheduled follow up visit.

DETAILED DESCRIPTION:
In order to perform a patient specific ACL reconstruction we have developed a surgical instrument (SONAR femoral Aimer PSI) that can be used during an outside-in ACL reconstruction.

The SONAR femoral Aimer PSI is an adaption to the RetroConstruction™ Guide, type AR-1510 used in the GraftLink® technique. This technique is now used in approximately 70% of ACL reconstructions in the Netherlands (information supplied by Arthrex).

In the SONAR femoral Aimer PSI the tip of the guide is designed for each individual patient based on the pre-operative MRI. In the 3D laboratory from the UMCG, the images from the MRI are loaded in a software program used for digital image processing called Mimics.

Using Mimics, the bone and cartilage of the distal femur are segmented, which is a digital method to create a 3D model of the distal femur and overlying cartilage.

Based on this 3D model, a negative mold is created which fits the intercondylar notch of the knee. This patient specific design is transferred to the Research Instrument Manufactory (RIM) of the UMCG. At the RIM a computerized cutter with 6 degrees of freedom is used to create the SONAR femoral aimer PSI from stainless steel.

After proper sterilisation of the instrument, as described in appendix 2, the instrument is ready to be used during a patient specific ACL reconstruction.

The SONAR femoral Aimer PSI has been used in cadaver experiments and had led to a mean deviation of 3.0 mm when based on a 2D MRI .

The aim of this study is to determine the in vivo accuracy of the SONAR Femoral Aimer PSI. and to monitor general safety aspects.

Subjects will undergo ACL reconstruction in which the Femoral Aimer PSI will be used for femoral tunnel positioning. Both pre- and postoperative care will be provided as usual.

At all times during the intervention it is possible for the surgeon to " fall back" on the usual care technique of ACL reconstruction.

Subjects are not exposed to other risks than those accompanying routine ACL reconstruction.

Subjects can leave the study at any time for any reason if they wish to do so without any consequences. The investigator can decide to withdraw a subject from the study for urgent medical reasons.

The treating surgeon can decide to withdraw a subject from the study during surgery if the SONAR Femoral Aimer PSI does not lead to a satisfactory tunnel position. This decision is based on the experience of the treating surgeon and cannot be disputed by the sponsor or members of the research team.

After withdrawal of a subject, subjects will be replaced to reach a study population of 10 subjects.

In accordance to section 10, subsection 4, of the WMO, the sponsor will suspend the study if there is sufficient ground that continuation of the study will jeopardise subject health or safety. The sponsor will notify the accredited METC without undue delay of a temporary halt including the reason for such an action. The study will be suspended pending a further positive decision by the accredited METC. The investigator will take care that all subjects are kept informed.

Adverse events are defined as any undesirable experience occurring to a subject during the study, whether or not considered related to the investigational product. All adverse events reported spontaneously by the subject or observed by the investiga¬tor or his staff will be recorded.

A serious adverse event is any untoward medical occurrence or effect that

* results in death;
* is life threatening (at the time of the event);
* requires hospitalisation or prolongation of existing inpatients' hospitalisation;
* results in persistent or significant disability or incapacity;
* is a congenital anomaly or birth defect; or
* any other important medical event that did not result in any of the outcomes listed above due to medical or surgical intervention but could have been based upon appropriate judgement by the investigator.

An elective hospital admission will not be considered as a serious adverse event.

The investigator will report all SAEs to the sponsor without undue delay after obtaining knowledge of the events.

The sponsor will report the SAEs through the web portal ToetsingOnline to the accredited METC that approved the protocol, within 7 days of first knowledge for SAEs that result in death or are life threatening followed by a period of maximum of 8 days to complete the initial preliminary report. All other SAEs will be reported within a period of maximum 15 days after the sponsor has first knowledge of the serious adverse events.

In addition to the expedited reporting of SUSARs, the sponsor will submit, once a year throughout the clinical trial, a safety report to the accredited METC, competent authority, and competent authorities of the concerned Member States.

This safety report consists of:

* a list of all suspected (unexpected or expected) serious adverse reactions, along with an aggregated summary table of all reported serious adverse reactions, ordered by organ system, per study;
* a report concerning the safety of the subjects, consisting of a complete safety analysis and an evaluation of the balance between the efficacy and the harmfulness of the medicine under investigation.

All AEs will be followed until they have abated, or until a stable situation has been reached. Depending on the event, follow up may require additional tests or medical procedures as indicated, and/or referral to the general physician or a medical specialist.

SAEs need to be reported till end of study within the Netherlands, as defined in the protocol

A Data Safety Monitoring Board (DSMB) or Safety Committee will not be installed.

A structured risk analysis has been performed. Based on the outcome of the structured risk analysis, a monitor will be selected from the UMCG monitor pool to monitor the study.

The study will be conducted according to the principles of the Declaration of Helsinki (version 9, oct 2008 Seoul), See for the most recent version: www.wma.net).

Subject will be recruited by their treating orthopaedic surgeon when they are enlisted for ACL reconstruction surgery. Subjects will receive oral and written information concerning the study. Subjects are asked to provide written informed consent within two weeks after their visit.

An independent expert is available for subjects. Subjects can address this expert if they wish to discuss study matters with an independent person, not linked to the study.

Contact details will be given in patient information letters.

The sponsor/investigator has a liability insurance which is in accordance with article 7 of the WMO.

The sponsor (also) has an insurance which is in accordance with the legal requirements in the Netherlands (Article 7 WMO). This insurance provides cover for damage to research subjects through injury or death caused by the study.

The insurance applies to the damage that becomes apparent during the study or within 4 years after the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* >16 years
* Primary ACL injury requiring ACL reconstruction

Exclusion Criteria:

* No preoperative MRI available.
* Inability to understand the Dutch language (assessed by the treating physician)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy | 2 weeks post surgery
  Deviation in mm of realised femoral tunnel position compared to planned femoral tunnel position. Measured on pre and postoperative MRI

SECONDARY OUTCOMES:
Complications | 2 weeks post surgery
  The occurence of per and postoperative complications

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Ommelander Ziekenhuis Groningen, Scheemda, Provincie Groningen
  - University Medical Centre Groningen, Groningen

IPD SHARING:
Plan to Share IPD: Undecided